CLINICAL TRIAL: NCT04725409
Title: Neural Correlates of Neuropsychiatric Functions
Brief Title: Neural Correlates of Psychiatric Disorders
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Bick, Assistant Professor of Neurosurgery, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 211037
Record Dates: First submitted 2021-01-14; First posted 2021-01-26 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Psychiatric Disorder; Memory Disorders
Keywords: Depression; Stereo Electroencephalography (SEEG); Anxiety; Obsessive compulsive disorder; Impulsivity; Memory
MeSH Terms: conditions — Mental Disorders; Memory Disorders; Depression; Anxiety Disorders; Obsessive-Compulsive Disorder; Impulsive Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — EEG recordings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Epilepsy patients: All participants will be patients with medically refractory epilepsy undergoing depth electrode placement for seizure localization. For this study, participants will complete psychiatric questionnaires measuring depression, anxiety, obsessive compulsive disorder, and impulsivity, and EEG recordings will be collected from the depth electrodes while subjects rest quietly. Some subjects will also participate in neuro cognitive tasks while neural recordings/stimulation are performed. Some subjects will also undergo macro-micro electrode implantation as a part of their SEEG implantation procedure for the purpose of EEG macro (local activity) and micro (single-unit) recordings.

SUMMARY:
This ClincialTrials.gov record originally corresponded to the protocol approved under IRB # 202370. The study was expanded to include stimulation and recordings approved under new IRB #211037. The participant data originally acquired from IRB# 202370 will be included in this new record:

This study seeks to better understand the neural activity underlying neuro cognitive disorders. Resting state local field potential recordings will be collected from medically refractory epilepsy patients implanted with depth electrodes for seizure localization, and metrics of neural activity will be correlated with psychiatric symptoms as measured from questionnaires. Subjects will also participate in neuro cognitive tasks while neural recordings are performed, and/or receive neural stimulation through implanted depth electrodes. A better understanding of disordered neural activity underlying neuropsychiatric disorders may additionally contribute to novel methods for diagnosing, treating, and preventing these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing SEEG monitoring at Vanderbilt University Medical Center
* At least 18 years of age
* English speaking

Exclusion Criteria:

* Age <18
* Not able to complete questionnaires (e.g., unable to comprehend instructions or follow directions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with medically refractory epilepsy who have undergone depth electrode placement for localization of their refractory seizures.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Neural activity correlating with the Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) | During patient's epilepsy monitoring stay, approximately 15 minutes
  The Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) is a commonly used and well validated depression screening tool consisting of 20 questions. Scores range from 0 to 60 and a score of 16 or above indicates a risk for clinical depression. CESD-R scores will be correlated with resting state measures of neural activity and connectivity
Neural activity correlating with the State-Trait Anxiety Inventory (STAI) | During patient's epilepsy monitoring stay, approximately 15 minutes
  The State-Trait Anxiety Inventory (STAI) is a validated anxiety scale that screens for current anxiety state and chronic anxiety trait. It consists of 40 questions with scores ranging from 20 to 80. A score of 40 or above indicates risk of anxiety. STAI scores will be correlated with resting state measures of neural activity and connectivity
Neural activity correlating with the Yale-Brown Obsessive Compulsive Scale (YBOCS) | During patient's epilepsy monitoring stay, approximately 15 minutes
  The Yale-Brown Obsessive Compulsive Scale (YBOCS) is the most commonly used and well validated measure of obsessive compulsive features. It consists of 10 questions with scores ranging from 0 to 40. A score of 8-15 indicates mild OCD, 16-23 indicates moderate OCD, 24-31 indicates severe OCD and 32-40 indicates extreme OCD. YBOCS scores will be correlated with resting state measures of neural activity and connectivity
Neural activity correlating with the Barratt Impulsiveness Scale (BIS11) | During patient's epilepsy monitoring stay, approximately 15 minutes
  The Barratt Impulsiveness Scale (BIS11) is a well validated measure of impulsive traits that consists of 30 questions. The scores of the BIS11 range from 30 to 120 with scores above 72 indicating high levels of impulsivity. BIS11 scores will be correlated with resting state measures of neural activity and connectivity
Local field potential changes in response to study tasks | During patient's epilepsy monitoring stay, approximately 20-30 minutes
  These local field potential changes are neural recordings in response to the stop signal tasks and n back tasks. In the stop signal reaction time task the subject will see a visual stimulus and be asked to press a button to respond. On some trials an auditory stimulus will also be presented which will indicate that the subject should not press the response button (they should suppress their response). In the n-back verbal working memory task the subject will see a series of words presented sequentially on a screen. During each word presentation the subject will press a button to indicate whether or not the word matches that presented n trials prior
Behavioral performance changes with stimulation | During patient's epilepsy monitoring stay, approximately 20-30 minutes
  Stimulation will occur during the stop signal task and n back task. In the stop signal reaction time task the subject will see a visual stimulus and be asked to press a button to respond. On some trials an auditory stimulus will also be presented which will indicate that the subject should not press the response button (they should suppress their response). In the n-back verbal working memory task the subject will see a series of words presented sequentially on a screen. During each word presentation the subject will press a button to indicate whether or not the word matches that presented n trials prior. Stimulation will be delivered through pre-selected SEEG electrodes via the Ripple Neuromed Summit system. Test stimulation will be performed prior to stimulation during the task to test for safety and tolerability, with the patient monitored for symptoms by a neurosurgeon or neurologist.
Single unit neuronal spiking changes in response to study tasks | During patient's epilepsy monitoring stay, approximately 20-30 minutes
  Single neuron (single unit) spiking activity is recorded through SEEG micro neural recordings in response to patients completing neuro cognitive tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bick, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No